CLINICAL TRIAL: NCT06588777
Title: Ultrasound Guided Modified Thoracoabdominal Nerve Block Through Perichondrial Approach (M-TAPA) Versus Quadratus Lumborum Block for Postoperative Analgesia in Laparoscopic Cholecystectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Hassan Helmy, Clinical Doctor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MD92/2024
Record Dates: First submitted 2024-09-01; First posted 2024-09-19 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Laparoscopic Cholecystectomy; Modified Thoracoabdominal Nerve Block; Quadratus Lumborum Block
Keywords: Laparoscopic cholecystectomy; modified thoracoabdominal nerve block; quadratus lumborum block

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified thoracoabdominal nerve block through perichondrial approach (M-TAPA) (Experimental): Using the in plane technique A deep angle was given to the costochondral angle at the edge of the 10th costal margin with the probe in the sagittal direction to view the lower surface of the costal cartilage in the midline. A 22-G, 100-mm block needle will be inserted in the cranial direction using the in-plane technique and the needle tip will be moved to the posterior aspect of the 10th costal cartilage. It is noted that the needle tip never crossed the cranial edge of the 10th costal cartilage and 20 mL of 0.25% bupivacaine will be injected into the lower surface of the chondrium to make Modified thoracoabdominal nerve block through perichondrial approach (M-TAPA).
  Interventions: Procedure: Modified thoracoabdominal nerve block through perichondrial approach (M-TAPA)
- Quadratus lumborum block (Experimental): Using the in plane technique the probe will be placed in the mid-axillary line between the lower costal margin and the iliac crest in a transverse plane to view all abdominal layers. The probe will be moved towards the posterior axillary line, to reach a point where all three abdominal muscle layers merge to form aponeurosis.
  The aponeurosis will then be followed dorsally until the quadratus lumborum muscle is seen deep to transversalis fascia with its attachment to the transverse process of the L4 vertebral body. A 22 G, 100 mm, blunt, insulated nerve block needle will be inserted 1 cm medial to the probe and advanced using the in-plane technique with ultrasound real-time assessment. The injection site will be the junction of transversalis fascia and the anterolateral border of quadratus lumborum muscle.
  Interventions: Procedure: Quadratus lumborum block

INTERVENTIONS:
Procedure: Modified thoracoabdominal nerve block through perichondrial approach (M-TAPA) — transversus abdominis, internal oblique, and external oblique muscles will be identified with a high-frequency (10 MHz) linear probe on the costochondral angle in the sagittal plane under ultrasound guidance at the 10th costal margin. A deep angle was given to the costochondral angle at the edge of the 10th costal margin with the probe in the sagittal direction to view the lower surface of the costal cartilage in the midline. A 22-G, 100-mm block needle will be inserted in the cranial direction using the in-plane technique and the needle tip will be moved to the posterior aspect of the 10th costal cartilage. It is noted that the needle tip never crossed the cranial edge of the 10th costal cartilage
  Other Names: (M-TAPA)
  Arms: Modified thoracoabdominal nerve block through perichondrial approach (M-TAPA)
Procedure: Quadratus lumborum block — using ultrasound guidance (Sonosite turbo M, Bothell, Washington, USA) and a curved ultrasound probe (2.5-7.5 MHz). The probe will be placed in the mid-axillary line between the lower costal margin and the iliac crest in a transverse plane to view all abdominal layers. The probe will be moved towards the posterior axillary line, to reach a point where all three abdominal muscle layers merge to form aponeurosis.
  The aponeurosis will then be followed dorsally until the quadratus lumborum muscle is seen deep to transversalis fascia with its attachment to the transverse process of the L4 vertebral body. A 22 G, 100 mm, blunt, insulated nerve block needle will be inserted 1 cm medial to the probe and advanced using the in-plane technique with ultrasound real-time assessment. The injection site will be the junction of transversalis fascia and the anterolateral border of quadratus lumborum muscle
  Other Names: (QLB)
  Arms: Quadratus lumborum block

SUMMARY:
This study aims to compare the efficacy of using Ultrasound guided modified thoracoabdominal nerve block through perichondrial approach (M-TAPA) versus quadratus lumborum block for postoperative analgesia in laparoscopic cholecystectomy under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aging ≥ 21 years to ≤ 70 of both sexes.
* Patients undergoing Laparoscopic cholecystectomy surgeries.
* ASA physical status classes I - II.

Exclusion Criteria:

* Patient's refusal of procedure or participation in the study.
* ASA classes III or above.
* Coagulopathy and bleeding disorders.
* Evidence of Local skin infections at site of injection.
* Body mass index >40kg/m2
* A history of relevant local anesthetic allergy.

Ages: 21 Years to 71 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Time to first Rescue Analgesia | 24 hours postoperative
  Is to measure the first time to resque analgesia postoperative (24 hours)

SECONDARY OUTCOMES:
The total requirements of rescue analgesia Meperidine (pethidine) over the first 24 hours postoperative | 24 hours postoperative
Heart rate | at intervals of 0 (PACU), 1, 2, 4, 6, 12, 18 and 24 hours postoperatively
Blood pressure | at intervals of 0 (PACU), 1, 2, 4, 6, 12, 18 and 24 hours postoperatively
Spo2 measuring | at intervals of 0 (PACU), 1, 2, 4, 6, 12, 18 and 24 hours postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Ainshams university hospitals, Cairo, Egypt